CLINICAL TRIAL: NCT04196075
Title: The Effect of Andrographis Paniculata (AP) on Palliative Management of Advanced Esophageal Cancer
Acronym: AP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Philip Wai Yan CHIU, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CRE-2017.616
Record Dates: First submitted 2019-12-10; First posted 2019-12-12 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Squamous Cell Carcinoma of Esophagus
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Andrographis paniculata extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Andrographis Paniculata treatment (Experimental): Single lot of Andrographis paniculata (AP) concentrated granules (Andrographis Herba) will be manufactured by Nong's Company Limited under GMP standard
  Interventions: Drug: Andrographis Paniculata

INTERVENTIONS:
Drug: Andrographis Paniculata — AP as palliative treatment

SUMMARY:
This is a prospective cohort study on the effect of Andrographis Paniculata (AP) on palliative management of patients with advanced or metastatic esophageal cancer. A total of 30 patients with locally advanced or metastatic squamous esophageal cancer will be recruited for the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged over 18
2. Locally advanced esophageal cancer with invasion or adherent to surrounding organs including trachea, recurrent laryngeal nerves and descending aorta;
3. Presence of distant metastasis;
4. Extensive lymph node metastasis to beyond surgical therapy

Exclusion Criteria:

1. Patients who cannot receive palliative stenting for dysphagia or under other conventional treatment including chemotherapy or chemoradiotherapy
2. Patients who are not willing to receive Chinese herbal medicines
3. Patients who do not consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Symptomatic relief and quality of life after AP | 4 months
  Symptomatic relief of Dysphagia and quality of life after treatment Dysphagia measured by Dysphagia score Quality of Life measured by EORTC-QLQ-C30

SECONDARY OUTCOMES:
Difficulty to swallow | 4 months
  Difficulty to swallow by dysphagia grade 0 = able to eat normal diet / no dysphagia.
  1. = able to swallow some solid foods
  2. = able to swallow only semi solid foods
  3. = able to swallow liquids only
  4. = unable to swallow anything / total dysphagia
Survival | up to 36 months
  Median Survival
Adverse events | up to 36 months
  Rate of adverse events
AP side effects | 4 months
  Side effects related to AP including
  1. Gastrointestinal upset
  2. Nausea and Vomiting
  3. Allergy
  4. Diarrhoea
  5. Abdominal pain
  6. Dizziness

CONTACTS AND LOCATIONS:
Overall Officials: Philip WY Chiu, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Surgery, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong, Outside of US & Canada, China

IPD SHARING:
Plan to Share IPD: Undecided